CLINICAL TRIAL: NCT01295814
Title: An Investigator Initiated, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy of Humira® (Adalimumab) For The Treatment of Interstitial Cystitis(IC)
Brief Title: Efficacy Study of Adalimumab to Treat Interstitial Cystitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ICStudy, LLC (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Philip C. Bosch, M.D., Urologist, ICStudy, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMM 10-0061
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial cystitis; Humira; Adalimumab
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adalimumab (Experimental): Adalimumab 80mg subcutaneous loading dose followed by 40 mg subcutaneous every 2 weeks for 12 weeks
  Interventions: Drug: Adalimumab
- Inactive drug (Placebo Comparator): Placebo in identical syringe subcutaneous every 2 weeks for 12 weeks
  Interventions: Other: inactive drug

INTERVENTIONS:
Drug: Adalimumab — 80 mg loading dose given subcutaneously followed by 40 mg dose given subcutaneously every two weeks over a twelve week period
  Other Names: Humira
  Arms: adalimumab
Other: inactive drug — 80 mg loading dose given subcutaneously followed by 40 mg dose given subcutaneously every two weeks over a twelve week period
  Other Names: placebo
  Arms: Inactive drug

SUMMARY:
The purpose of this study is to evaluate an investigational treatment for interstitial cystitis. Interstitial cystitis is a chronic bladder disease that includes the following symptoms: Urinary frequency during the day,urinary frequency at night, urinary urgency and bladder discomfort relieved by voiding.

Presently, there is no cure for interstitial cystitis. The response to current treatments is poor. Patients with interstitial cystitis have a poorer quality of life. The cause of interstitial cystitis is unknown. This study is evaluating the drug Humira® (adalimumab) for improving the symptoms of patients with interstitial cystitis. Humira® is an injectable anti-inflammatory medication that has been available for use since December 31, 2002. Humira® has been FDA approved for the treatment of rheumatoid arthritis, psoriasis, ankylosing spondylitis, and Crohn's disease. These diseases have similar characteristics to interstitial cystitis. This study will evaluate an investigational use of Humira® for the treatment of interstitial cystitis.

DETAILED DESCRIPTION:
Interstitial cystitis (IC) is a chronic disabling bladder syndrome characterized by urinary frequency, nocturia, urinary urgency, and pain with bladder filling-relieved by emptying. There is no cure for IC and the treatment options are suboptimal. Patients with IC report significant negative effects on their physical and mental quality of life. The etiology of IC is unknown. Certain aspects of IC suggest that autoimmunity may play a role in initiating or sustaining the chronic inflammatory response. Bladder biopsies of patients with IC demonstrate an increase number of mast cells. Mast cell activation with the release of tumor necrosis factor (TNF) may mediate this bladder inflammation. Humira® (adalimumab) is a medication that blocks the effect of TNF. Humira® (adalimumab) is FDA approved for the treatment of rheumatoid arthritis, psoriasis, ankylosing spondylitis, and Crohn's disease. These diseases are similar to IC. In this study, the hypothesis being tested is that Humira® (adalimumab) will show efficacy at reducing the symptoms of IC.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥18 and ≤ 65 years of age previously diagnosed with Interstitial Cystitis
* Currently have symptoms of urinary urgency, frequency or pain for more than 6 months
* Urinating at least 7 times a day or having some urgency or pain (measured on linear analog scales)
* Must be post-menopausal or surgically sterile or willing to use an adequate form of birth control
* Not pregnant or lactating
* Capable of voiding independently
* Willing to provide informed consent to participate

Exclusion Criteria:

* Have symptoms that are presently relieved on other medications for interstitial cystitis
* Have absence of nocturia
* Have symptoms that are relieved by antimicrobials or antibiotics.
* Have a body mass index (BMI) of >39 kg/m2
* Have uncontrolled hypertension
* Have Type I or type 2 diabetes
* Have active Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV) infection, or who are known carriers (Hepatitis B) at Screening
* Have a positive tuberculosis test at screening
* Have had a urinary tract infection for 6 weeks
* Have had bacterial cystitis in previous 3 months
* Have had previous exposure to Humira® (adalimumab)
* Have taken investigational medication within 30 days of screening
* Have any other condition/disease which, in the opinion of the investigator, could compromise subject safety or confound the interpretation of study results
* Are unable or unwilling to comply with protocol requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Bosch, MD, Principal Investigator
Locations (1):
- Philip C. Bosch, MD, Escondido, California, United States

REFERENCES:
- [Result] Bosch PC. A randomized, double-blind, placebo controlled trial of adalimumab for interstitial cystitis/bladder pain syndrome. J Urol. 2014 Jan;191(1):77-82. doi: 10.1016/j.juro.2013.06.038. Epub 2013 Jun 20. PMID 23792149
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subject were recruited from medical practices and by advertisement starting March 2011 through January 2013.
Pre-assignment Details: A total of 4 subjects did not meet screening criteria.
Groups:
- Inactive Drug: inactive drug : placebo
- Adalimumab: Adalimumab : 80 mg loading dose given subcutaneously followed by 40 mg dose given subcutaneously every two weeks over a twelve week period
Period: Overall Study
Arm/Group | Inactive Drug | Adalimumab
Started | 22 | 21
Completed | 20 | 19
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactive Drug | Adalimumab | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (13.4) | 45.2 (14) | 45.9 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: O'Leary-Santa Interstitial Cystitis Symptom Index and Problem Index (OSPI) Score
Description: Improvement in the O'Leary Sant Symptom and Problem Index from baseline to week 12 Total scores on a scale range: 0-36 (0, meaning no symptoms to 36, meaning the most severe symptoms)
Time Frame: Baseline/12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inactive Drug | Adalimumab
Number analyzed (Participants) | 22 | 21
units on a scale
  Baseline | 27.7 (4.9) | 27.8 (3.9)
  Week 12 | 19.6 (10.7) | 19.9 (7.5)
Statistical Analysis 1: Comparison: Inactive Drug vs Adalimumab; Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Test type: Non-Inferiority or Equivalence — The study had acceptable sensitivity with a statistical power of 0.99 (99%) for the improvement in the adalimumab group from baseline to week 12. The study had acceptable sensitivity with a statistical power of 0.92 (92%) for the improvement in the placebo group from baseline to week 12; p = 0.75, t-test, 2 sided — Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Mean Difference (Final Values) = 7.9, 95% CI 2-sided [4.0 to 11.8] — Confidence interval was improvement in OSPI in the adalimumab group from baseline to week 12

2. Secondary Outcome: Interstitial Cystitis Symptom Index (ICSI)
Description: Improvement in O'Leary Sant Interstitial Cystitis Symptom Index (ICSI) Total scores on a range scale: 0-20 (0, meaning no symptoms, to 20, meaning the most severe symptoms)
Time Frame: Baseline/ 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inactive Drug | Adalimumab
Number analyzed (Participants) | 22 | 21
units on a scale
  Baseline | 14.2 (3.1) | 14.0 (2.7)
  Week 12 | 10.5 (5.7) | 10.0 (4.2)
Statistical Analysis 1: Comparison: Inactive Drug vs Adalimumab; Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Test type: Superiority or Other; p = 0.99, t-test, 2 sided — Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [1.7 to 6.3] — Confidence interval was improvement in ICSI in the adalimumab group from baseline to week 12

3. Secondary Outcome: Interstitial Cystitis Problem Index (ICPI)
Description: Improvement in O'Leary Sant Interstitial Cystitis Problem Index (ICPI) Total scores on a scale: 0-16 (0, meaning no symptoms, to 16, meaning the most severe symptoms)
Time Frame: Baseline/12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inactive Drug | Adalimumab
Number analyzed (Participants) | 22 | 21
units on a scale
  Baseline | 13.5 (2.2) | 13.8 (1.7)
  Week 12 | 9.1 (5.1) | 9.9 (3.6)
Statistical Analysis 1: Comparison: Inactive Drug vs Adalimumab; Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Test type: Superiority or Other; p = 0.76, t-test, 2 sided — Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [2.1 to 5.8] — Confidence interval was improvement in ICPI in the adalimumab group from baseline to week 12

4. Secondary Outcome: Pelvic Pain Urgency/Frequency (PUF) Score
Description: Pelvic Pain, Urgency/Frequency Symptom Scale Total scores on a scale range: 0-35 (0, meaning no symptoms, to 35, meaning the most severe symptoms)
Time Frame: Baseline12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inactive Drug | Adalimumab
Number analyzed (Participants) | 22 | 21
units on a scale
  Baseline | 24.2 (3.9) | 24.6 (4.1)
  Week 12 | 17.3 (8.7) | 18.3 (6.9)
Statistical Analysis 1: Comparison: Inactive Drug vs Adalimumab; Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Test type: Superiority or Other; p = 0.76, t-test, 2 sided — Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [2.6 to 10.0] — Confidence interval was improvement in PUF in the adalimumab group from baseline to week 12

5. Secondary Outcome: Global Response Assessment (GRA)
Description: Percent(%) of patients who reported 50% or greater overall improvement in their condition.
  Score on a scale range (improvement 0%-100%)
Time Frame: Measured at12 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Inactive Drug | Adalimumab
Number analyzed (Participants) | 22 | 21
percentage of participants | 50 | 53
Statistical Analysis 1: Comparison: Inactive Drug vs Adalimumab; Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12; Test type: Superiority or Other; p = 0.67, t-test, 2 sided — Statistical improvement in the adalimumab group compared to the placebo group from baseline to week 12

ADVERSE EVENTS:
Time Frame: 2 years
Description: March 2011 to March 2013
Arm/Group | Inactive Drug | Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 21/22 | 17/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inactive Drug (N=22) | Adalimumab (N=21)
Diarrhea (Gastrointestinal disorders) | 7 (8) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (10)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 12 (14)
Pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 3 (3) — Does not include headache
Headache (General disorders) | 5 (10) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3) | 5 (8)
Salmonella (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dizziness (General disorders) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other